CLINICAL TRIAL: NCT07189520
Title: SAFE-AI ONCO-TRACK: Multimodal GenAI for Early Detection of Minimal Residual Disease and Recurrence in Gastrointestinal Oncology
Brief Title: 1. SAFE-AI ONCO-TRACK: Multimodal GenAI for Early Detection of Minimal Residual Disease and Recurrence in Gastrointestinal Oncology
Acronym: ONCO-TRACK
Status: Not yet recruiting | Type: Observational
Sponsor: Università Politecnica delle Marche (Other)
Responsible Party: Principal Investigator, Monica Ortenzi, Assistant Professor, Università Politecnica delle Marche
Other Study IDs: SAFE-AI ONCO-TRACK; 2025-TOOL-01-03 (Other: Università Politecnica delle Marche)
Record Dates: First submitted 2025-09-16; First posted 2025-09-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — Artificial Intelligence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — consistent prognostic value for minimal residual disease (MRD) and recurrence risk. However, most available studies are heterogeneous in assays, sampling timepoints, and outcome definitions, and are predominantly retrospective or single-centre, which limits their generalizability and clinical utility.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- AI cohort: Benchmark AI scoring vs expert raters (GEARS/OCHRA κ ≥0.75)• Assess performance gains after GenAI feedback (≥15% improvement)• Measure usability, cognitive load, and ecological footprint reduction
  Interventions: Other: Artificial Intelligence

INTERVENTIONS:
Other: Artificial Intelligence — Benchmark AI scoring vs expert raters (GEARS/OCHRA κ ≥0.75)• Assess performance gains after GenAI feedback (≥15% improvement)• Measure usability, cognitive load, and ecological footprint reduction

SUMMARY:
Current decision tools (TNM, MRI/PET, CEA, and other serum markers, as well as single-marker genomics) are insufficiently predictive of responders, fail to detect early MRD in many cases, and rarely connect molecular biology to dynamic perioperative data. SAFE-AI will build and validate multimodal, explainable GenAI models that fuse liquid/tissue multi-omics with radiology and clinical trajectories to:

(i) detect MRD earlier, (ii) improve recurrence-risk calibration, and (iii) support non-invasive "virtual biopsy"-inferring tissue-level features from blood profiles, and vice-versa, to mitigate missing-modality gaps. This is grounded in the strong mechanistic premise that integrating heterogeneous molecular signals with imaging captures tumour-host biology more completely than single-modality assays, enabling actionable, calibrated risk estimates for rectal and oesophageal cancer.

The clinical hypothesis is that such integrated models can improve recurrence prediction by at least 20% over guideline baselines, with transparent uncertainty and bias monitoring to meet EU AI Act/MDR expectations.

DETAILED DESCRIPTION:
Current decision tools (TNM, MRI/PET, CEA, and other serum markers, as well as single-marker genomics) are insufficiently predictive of responders, fail to detect early MRD in many cases, and rarely connect molecular biology to dynamic perioperative data. SAFE-AI will build and validate multimodal, explainable GenAI models that fuse liquid/tissue multi-omics with radiology and clinical trajectories to:

(i) detect MRD earlier, (ii) improve recurrence-risk calibration, and (iii) support non-invasive "virtual biopsy"-inferring tissue-level features from blood profiles, and vice-versa, to mitigate missing-modality gaps. This is grounded in the strong mechanistic premise that integrating heterogeneous molecular signals with imaging captures tumour-host biology more completely than single-modality assays, enabling actionable, calibrated risk estimates for rectal and oesophageal cancer.

The clinical hypothesis is that such integrated models can improve recurrence prediction by at least 20% over guideline baselines, with transparent uncertainty and bias monitoring to meet EU AI Act/MDR expectations.

ELIGIBILITY:
Inclusion Criteria (Justification in parenthesis):

* Age ≥18 years (RC and EC are primarily adult-onset cancers, and adult inclusion aligns with ethical biospecimen collection and consent processes.)
* Histologically confirmed diagnosis of rectal or esophageal cancer (Confirms clinical relevance and eligibility for standard treatment pathways.)
* Treatment plan includes surgical resection with curative intent (Ensures applicability to MRD and outcome prediction tasks.)
* Undergoing standard-of-care neo-adjuvant or perioperative therapy (Ensures data consistency and relevance to response modelling.)
* Ability and willingness to provide informed consent for biospecimen and clinical data use (Meets ethical requirements for participation.)
* Availability for longitudinal blood sampling at T0 (baseline), T1 (3 months post-treatment), and T2 (6 months post-treatment) (Critical for temporal biomarker analysis.)
* Optional Inclusion: Access to tumor tissue (archival or fresh) for multi-omic profiling (Supports deep integrative biomarker discovery.)

Exclusion Criteria:

* Diagnosis of non-resectable or metastatic disease at enrollment (Excludes non-curative settings where the longitudinal biomarker protocol may not be feasible.)
* Emergency surgeries or treatment plans that deviate from standard protocols (To maintain data comparability.)
* Inability or refusal to provide informed consent (Essential for ethical compliance.)
* Failure to complete biospecimen donation or key follow-up timepoints (Maintains data integrity and model reliability.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2028-06-01 (Estimated); Study Completion 2030-06-01 (Estimated)

PRIMARY OUTCOMES:
Primary outcomes | 24 months
  Primary Objective A: Establish a generative AI-powered simulation ecosystem (SAFE-AI) for biomarker discovery, risk stratification, and safety testing in oncology through integration of synthetic data, 3D tumour models, and multi-omics datasets. (Threshold: AUC ≥0.80 (95% CI ±0.05) for 12-mo recurrence prediction; Model calibration slope ≥0.90)